CLINICAL TRIAL: NCT07017881
Title: The Effect of Psychosocial Skills Training Applied to Individuals Diagnosed With Schizophrenia on Subjective Recovery, Self-Esteem and Quality of Life Levels
Brief Title: The Effectiveness of Psychosocial Skills Training Applied to Individuals Diagnosed With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neslihan Lok (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Sponsor-Investigator, Neslihan Lok, Prof. Dr. Study Director, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SELCUKU-ANCANDAN-001
Record Dates: First submitted 2025-05-25; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Schizophenia Disorder; Psychiatric Nursing; Psychosocial Skills Training
Keywords: schizophenia disorder; psychiatric nursing; Psychosocial skills training; quality of life; self-esteem; Subjective improvement

STUDY DESIGN:
Intervention Model Description: The sample group was determined as 48 in total, 24 intervention and 24 control. Individuals were assigned to the intervention and control groups using the simple randomization method. The program was asked to randomly divide the files into two groups of 24 people each. The researcher randomly determined these two groups as the intervention (Set 1) and control (Set 2) groups. The 24 individuals constituting the intervention group were assigned to 3 separate groups of 8 people each (Group 1, Group 2, Group 3) using the block randomization method. In addition to their routine treatments, the intervention group received one session of psychosocial skills training per week. The control group continued their routine treatments.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No intervention was applied. They continued their routine outpatient clinic check-ups and treatments.
- intervention group (Experimental): The intervention group is a group of 24 schizophrenia patients who received 11 weeks of Psychosocial Skills Training.
  Interventions: Behavioral: Psychosocial Skills Training

INTERVENTIONS:
Behavioral: Psychosocial Skills Training — The 24-person intervention group was divided into three separate groups of 8 people (Group 1, Group 2, Group 3). Group 1 and Group 2 attended sessions on Tuesdays at different times, while Group 3 attended sessions on Thursdays. Psychosocial Skills Training consisted of eleven sessions in total, one session per week. Sessions lasted an average of 60 minutes for each group. In each session, 5-10 minute breaks were given for rest and eating and drinking, considering the attention span and fatigue of the patients. Psychosocial Skills Training was applied two days a week (Group 1-2: Tuesday, Group 3: Thursday) in order to ensure that the patients could get more benefit from the application.
  Arms: intervention group

SUMMARY:
This study was conducted to investigate the effects of Psychosocial Skills Training on subjective recovery, self-esteem and quality of life levels of schizophrenia patients. The research is a randomized controlled trial. The research was conducted with 48 schizophrenia patients (Experimental: 24, Control: 24) registered in the Mental Health and Diseases Outpatient Clinic of a hospital. Personal Information Form, Subjective Recovery Assessment Scale, Rosenberg Self-Esteem Scale, Quality of Life Scale for Schizophrenia Patients were used to collect data. Data were collected by the researcher using the self-reporting face-to-face interview method in the form of pre-test and post-test. Psychosocial Skills Training was applied to the patients in the experimental group, one session per week, two days a week for 11 weeks, while the patients in the control group did not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having been diagnosed with Schizophrenia for at least 6 months according to ICD-10,
* Being registered with Selçuk University Medical Faculty Hospital Mental Health and Diseases Polyclinic,
* Coming to polyclinic check-ups regularly,
* Using antipsychotic medication regularly,
* Being at least a primary school graduate,

Exclusion Criteria:

* • Having an organic mental disorder or mental retardation,

  * Having a visual or hearing impairment,
  * Participating in a program similar to the intervention to be implemented.
  * Not attending at least two sessions of Psychosocial Skills Training,
  * Having an exacerbation period/hospitalization and experiencing a physical discomfort at a level that prevents attending sessions during the program process,
  * Wanting to leave the study,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Subjective Improvement Total Score Average | 11 weeks from pre-test to end of training
  The scale is evaluated based on the total score and the total score varies between 17-85. Higher scores obtained from the scale indicate that the individual perceives himself/herself as better recovered.

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale Society Score Average | 11 weeks from pre-test to end of training
  The scale score varies between 0 and 6 points. A score between 0 and 1 indicates "high self-esteem", a score between 2 and 4 indicates "medium self-esteem", and a score between 5 and 6 indicates "low self-esteem".
Quality of Life Scale Total Score Average for Schizophrenia Patients | 11 weeks from pre-test to end of training
  High scores (5-6) obtained from the scale indicate high quality of life and good adaptation, while low scores (0-1) reflect low quality of life and poor adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan LÖK, Prof. Dr., Study Director — Selcuk University
Locations (1):
- Selcuk University Faculty of Medicine Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No